CLINICAL TRIAL: NCT01873820
Title: A Randomized, Double-blind, Crossover Study Comparing the Tolerance of Two Forms of Vitamin C in Acid Sensitive Adults
Brief Title: Tolerance of Two Forms of Vitamin C in Acid-sensitive Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NBTY, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry); Moyad, Mark MD MPH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 07EAHT
Record Dates: First submitted 2013-05-14; First posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-06

CONDITIONS: Tolerance
Keywords: Vitamin C; calcium ascorbate; ascorbic acid
MeSH Terms: interventions — calcium ascorbate; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calcium ascorbate -> ascorbic acid (Experimental)
  Interventions: Dietary Supplement: Calcium ascorbate; Dietary Supplement: Ascorbic acid
- Ascorbic acid -> calcium ascorbate (Experimental)
  Interventions: Dietary Supplement: Calcium ascorbate; Dietary Supplement: Ascorbic acid

INTERVENTIONS:
Dietary Supplement: Calcium ascorbate
Dietary Supplement: Ascorbic acid

SUMMARY:
The purpose of this study is to compare the tolerance of two forms of vitamin C in adults with sensitivity to acidic foods.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by laboratory results and medical history
* Females not of child bearing potential
* Self-reported sensitivity to acidic foods
* Agrees to consume a low vitamin C diet

Exclusion Criteria:

* Pregnant, breastfeeding, or planning to become pregnant during the trial
* Use of medications known to interact with vitamin C or cause epigastric effects
* Use of supplements containing containing vitamin C
* Duodenal ulcer or gastric ulcer, gastritis, hiatus hernia, or gastroesophageal reflux disease (GERD) within past 3 months
* Use of antacids and/or acid suppressors within 4 weeks of randomization
* History of irritable bowel syndrome and related disorders
* Alcohol use > 2 standard alcoholic drinks per day; alcohol or drug abuse within the past year
* History of cardiac disease within the past 6 months
* History of or current diagnosis of cancer
* Uncontrolled hypertension
* Unstable renal and/or liver disease
* History of kidney stones
* Unstable psychiatric disorder
* History of or current immunocompromise
* History of hemoglobinopathies
* Participation in another clinical research trial <30 days
* Abnormal liver function
* Serum creatinine > 1.5 x upper limit of normal (ULN)
* Anemia of any etiology
* Uncontrolled and/or untreated thyroid disorder
* BMI ≥ 35 kg/m2
* Unstable medications <30 days
* Allergy or sensitivity to test article ingredients
* Cognitively impaired and/or unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-03; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gastrointestinal Symptom Rating Scale at 5 and 10 days | 0, 5 and 10 days

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize, Inc, London, Ontario, Canada